CLINICAL TRIAL: NCT03393273
Title: Induction and Consolidation With Elotuzumab Before and After Peripheral Stem Cell Autologous Graft in Elderly Patients With Multiple Myeloma
Brief Title: Elotuzumab in Patients With Multiple Myeloma Before and After Peripheral Stem Cell Autologous Graft
Acronym: IFM2016-03
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision in accordance with the promotor
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170103; 2017-001446-10 (EudraCT Number)
Record Dates: First submitted 2017-12-07; First posted 2018-01-08 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
Keywords: Stem Cell autologous graft; Elotuzumab; Multiple myeloma; Elderly
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elotuzumab (Experimental): This is a single arm phase II trial to assess the Very Good Partial Response rate of a strategy involving autologous hematopoietic stem cell transplantation, after intensive treatment and followed by consolidation phase, with elotuzumab, dexamethasone, velcade, and thalidomide in elderly patients.
  Interventions: Drug: Elotuzumab

INTERVENTIONS:
Drug: Elotuzumab — * Induction 4 cycles of 28 days Elotuzumab IV, 10 mg/Kg, D1, 8, 15, 22 Dexamethasone PO, 40 mg/d, D1, 8, 15 Velcade® IV, 1,3 mg/m2/d, D1, 4, 8, 11 Thalidomide PO, 100 mg/d, D1 to 21
  * melphalan 140-200 mg/m2 one day followed by autologous hematopoietic stem cell transplantation
  * Consolidation 2 cycles of 28 days (2 to 3 months after autograft) Elotuzumab IV, 10 mg/Kg, D1, 8, 15 and 22 Dexamethasone PO, 40 mg/d, D1, 8 and 15 Velcade® IV, 1,3 mg/m2/d, D1, 4, 8, and 11 Thalidomide® PO, 100 mg/d, D1 to 21
  Other Names: Empliciti®

SUMMARY:
This is a multicenter, open-label phase II study, assessing the efficacy of elotuzumab in elderly patients with multiple myeloma undergoing peripheral stem cell autologous graft

DETAILED DESCRIPTION:
In patients of 65 years of age or older, intensive treatment (TI) with hematopoietic stem cell autologous graft (ASCH) is not considered as the gold standard. Nowadays, given the rise of new treatments, new studies assessing TI with ASCH in elderly, seem required. The association bortezomib (VEL) - thalidomide (THAL) - dexamethasone (DEX) is considered as the standard induction (Kumar, Flinn et al. 2012, Ludwig, Viterbo et al. 2013). However, more and more strategies with immunotherapies are developed. Furthermore, it looks encouraging to use several monoclonal antibodies at different clinical development levels. Thus, elotuzumab (ELO) is an IgG1 (immunoglobulin gamma-1) (IgGκ) humanized monoclonal antibody directed against SLAMF7. SLAMF7 is a glycoprotein expressed by myeloma cells and natural killer (NK) but not by healthy tissues. Consequently, elotuzumab can kill specifically myeloma cells without affecting healthy tissues (Hsi, Steinle et al. 2008). A phase I study assessed the safety of ELO in association with VEL, REV (Lenalidomide) and DEX in induction first-line treatment in elderly patients with median age of 67 years (Usmani, Sexton et al. 2015). There were no significant increase of side effects with this association compared with side effects usually reported with VEL, REV and DEX. Thus, adding ELO could lead to an increase of response rate, with no increase of toxicity.

For more than 10 years, the standard intensive treatment associates a MEL (MELPHALAN) conditioning (200 mg/m2) with a blood graft. In a recent study, almost all patients aged between 65-69 and 70-74 years received MEL at 200 mg/m2. The adverse events rate was similar between the different ages and a very low non-tied relapse mortality. Thus, in elderly patients selected, the use of MEL at 200 mg/m2 seems sure.

Moreover, it's widely admitted that the conditioning treatment should be based on an efficient drugs association with a limited toxicity. Studies assessing consolidation treatment with an association of new drugs are limited. Initial results suggest that the use of new drugs after intensive treatment (IT) with ASCH should increase response rate and improve progression-free survival and global survival.

The aim of this study IFM 2016-03 is to assess intensive treatment (IT) with AHSCT (Autologous hematopoietic stem cell transplantation) in elderly and to associate the different steps (induction, high dose conditioning, consolidation) with immunotherapy. Given the prior results of IFM and international studies, a VGPR (Very Good Partial Response) rate of around 85% is expected.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma de novo.
* Stage DS (Durie-Salmon) : III, II, I with at least 1 symptomatic bone lesion (confirmed by radiology).
* Age > 65 years
* Indication for a first line treatment with induction, stem cell autologous graft and consolidation
* Available documentation including cytogenetic and International Staging System (ISS) of the initial diagnosis before inclusion,
* Effective contraceptive method for men with a partner of childbearing age during all the treatment period and within 6 months after the last cure
* Affiliated to social security
* Written informed consent
* Willingness and ability to respect the visits and all the demands required by the study
* Patient eligible to a high dose chemotherapy and fulfilling the following biological criteria :

  * Neutrophils ≥ 1,0 × 109/L
  * Platelets ≥ 75 ×109/L (platelets transfusions are not allowed within 3 days before inclusion)
  * Total bilirubin ≤ 1,5 × upper limit.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit
  * Creatinin clearance > 50 mL/min

Exclusion Criteria:

* Diagnosis and treatment for any other cancer within five years before inclusion or any diagnosis for any cancer. Patients with a skin cancer (except melanoma or carcinoma in situ) are not excluded in case of complete resection.
* Central nervous system disease
* Infection requiring an intravenous (IV) antibiotherapy or any severe infection within 14 days before inclusion
* Diagnosis of any of the following diseases : Waldenström disease, POEMS (polyneuropathy, endocrinopathy, organomegaly, monoclonal gammapathy and skin lesions), plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome or myeloproliferative disorder.
* Uncontrolled cardiopathy including : uncontrolled hypertension, uncontrolled heart arrhythmia, nonsymptomatic congestive cardiac failure, unstable angina or myocardial infarction within 6 months before inclusion
* Active infection with hepatitis B or C virus ; positive HIV serology
* Any comorbidity or severe concomitant disease incompatible with the patient inclusion or interfering with the safety assessment of the study treatments.
* Psychiatric history or any social condition limiting the patient compliance.
* Documented allergy to any studied treatment or any of their components.
* Disability to take oral treatments, inability or refusal to adhere to treatment constraints, or any digestive surgery interfering with oral absorption or treatment tolerance.
* Any experimental treatment within 30 days prior to the administration of the first dose of the studied treatmentParticipation to another clinical trial
* Prior participation to a clinical trial with elotuzumab, no matter the arm of treatment.
* Administration of any pharmaceutical speciality acting against myeloma - such as systemic corticosteroids (>10 mg of prednisone equivalent a day) or clarithromycin - within the month prior to the inclusion. In case of emergency, patients can receive dexamethasone (40mg/day, 4 consecutive days, maximum dose of 160mg) between screening and randomization

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Maximal response rate Assesment of the International Myeloma Working Group uniform response criteria | 1 month after the last consolidation cure
  Assesment of the International Myeloma Working Group uniform response criteria

SECONDARY OUTCOMES:
survival and progression-free survival | one year after the last consolidation cure
  Survival rate and global follow-up
  * Progression-free survival is defined as the duration between the beginning of treatment to the occurrence of a disease progression or death (whichever is the cause), according event occurring first.
  * Survival rate and global follow-up is defined as the duration between the start of treatment to death (whatever the cause).
evaluation of the answer to the treatment to improve or maintain the response | 12 month of treatment from inclusion
  Best response obtained or maintained for each therapeutical phase
Role of the consolidation phase in the improvement or maintenance of the response to the treatment Time before progression | From inclusion to month 36
  Time before progression
Conversion from negative residual disease to positive residual disease or maintenance of a negative residual disease during all therapeutical phases | from inclusion to month 36
  Conversion rate from negative residual disease to positive residual disease or maintenance of a negative residual disease during induction,intensive treatment (IT) with AHSC (autograft of hematopoietic stem cells) and consolidation
correlation between residual disease and duration of the response to the treatment | From inclusion to the end of the 12 treatment-month
  Comparison of response duration, overall survival and event-free survival between patients with negative residual disease and the other patients, after the induction phase and at the end of the treatment phase
Tolerance to each phase of treatment (the induction phase, the intensive treatment, the consolidation phase) | From inclusion to month 36
  Tolerance to each therapeutical phase will be assessed with:
  * ECOG (Eastern Cooperative Oncology Group) performance status
  * Adverse events rate, serious adverse events rate
  * Biological parameters (blood count and biochemistry)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hématologie et thérapie cellulaire, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided